CLINICAL TRIAL: NCT06469424
Title: An Active Surveillance, Post-Authorization Study to Characterize the Safety of Tofacitinib in Patients With Moderately to Severely Active Ulcerative Colitis in the Real-World Setting Using Data From the United Registries for Clinical Assessment and Research (UR-CARE) in the European Union (EU)
Acronym: PASS TOFA
Status: Recruiting | Type: Observational
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: PASS TOFA
Record Dates: First submitted 2024-06-07; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Ulcerative Colitis
Keywords: prospective observational study with medication
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1 (Tofacitinib cohort):: Initiation of tofacitinib (i.e., first ever prescription) from 01 July 2018 through to 31 March 2025
- Cohort 2 (Biologics cohort):: * Initiation (i.e., first ever prescription) of a specific biologic agent (any TNFi or non-TNFi agent) from 01 July 2018 through to 31 March 2025
  * No prior use of specific biologic agent prior to index date using all available data
- Cohort 3 (Immunosuppressants cohort):: * Initiation (i.e., first ever prescription) of a specific immunosuppressant agent (without concurrent biologic therapy) from 01 July 2018 through to 31 March 2025
  * No prior use of specific immunosuppressant prior to index date using all available data
- Cohort 4 (Naïve cohort):: * Patients diagnosed with UC since 01 July 2018 through to 31 March 2025
  * Patients with no history of surgery for UC (surgery suggests more severe disease, and such patients would not be representative of patients with generally mild disease in Cohort 4)

SUMMARY:
The purpose of this study is to estimate the incidence rates of malignancy, excluding non-melanoma skin cancer (NMSC), venous thromboembolic events VTE (deep venous thrombosis [DVT] and pulmonary embolism [PE]), NMSC, major adverse cardiac events (MACE), progressive multifocal leukoencephalopathy (PML), infections, hospitalization and specific antibiotic or antiviral treatment, lung cancer, lymphoma, herpes zoster, myocardial infarction (MI), gastrointestinal (GI) perforations, fractures, surgery for UC and death; through 4 sub-groups: adult patients with UC who initiate tofacitinib in the course of routine clinical care compared to other medications approved to treat UC.

DETAILED DESCRIPTION:
Rationale and background:

Tofacitinib, an inhibitor of the Janus kinase (JAK) family of kinases, was approved in the European Union (EU) in July 2018 at a dose of 5 mg twice daily or 10 mg twice daily for the treatment of adults with moderate-to-severe ulcerative colitis (UC), who have had an inadequate response, lost response, or were intolerant to either conventional therapy or a biologic agent. Malignancy excluding non-melanoma skin cancer (NMSC) is an important potential risk and venous thromboembolism (VTE) is an important identified risk associated with the use of tofacitinib, and follow-up of large cohorts of patients over a long period is needed to evaluate the risks of these safety events, as well as other potential safety events of interest, that may be associated with tofacitinib treatment. Pfizer will implement a post approval, active surveillance study of tofacitinib exposed and unexposed patients using actively collected prospective data included in the UR-CARE platform.

Research question:

What are the incidence rates of safety events of interest in adult patients with UC treated with tofacitinib in routine clinical care, as compared to the incidence rates in patients with UC treated with other approved systemic agents, and patients with UC naïve to biologics and immunomodulators/immunosuppressants (hereafter referred to as immunosuppressants)?

Study design:

This is an active cohort study of adult patients with UC aged ≥18 years treated with tofacitinib compared to patient receiving alternative treatment or not treatment. The study will use secondary data collected in the UR-CARE platform, which is an ongoing, prospective, observational, cohort of European Union (EU) patients with inflammatory bowel disease (IBD) with the primary aim of facilitating daily patient care and research studies in IBD. This study will focus only on patients with UC enrolled in the UR-CARE platform.

Variables:

The study variables include baseline patient characteristics (i.e., clinical and demographic characteristics, comorbidities, and current and past therapies), the primary outcomes of interest, and other safety events of interest.

Data sources:UR-CARE will be used as the only data source.

Study size:

This study is descriptive, and all eligible patients in UR-CARE registry during the study period who have consented to participate in the study will be included, with no upper limit on the sample size.

Data analysis:

All statistical analysis will be performed by GETECCU using SAS software v9.4, SAS Institute Inc, Cary, NC, USA. Detailed methodology for summary and statistical analyses of data collected in this study will be documented in a statistical analysis plan (SAP).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years,
* With Ulcerative colitis diagnosis per ECCO guidelines,
* Enrolled in UR-CARE registry with 12 months of medical history available in UR-CARE prior to the index date,
* With an informed consent signed. A minimum follow-up duration of 12 months will allow evaluation of safety events of interest.

Exclusion Criteria:

* Patients not meeting the inclusion criteria
* Patients who have any records of Crohn's Diseases (CD) or IBD unspecified in UR-CARE between the last UC diagnosis and index date [i.e. date of first prescription for tofacitinib].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with UC aged ≥18 years treated with tofacitinib compared to patient receiving alternative treatment or not treatment. The study will use secondary data collected in the UR-CARE platform, which is an ongoing, prospective, observational, cohort of European Union (EU) patients with inflammatory bowel disease (IBD) with the primary aim of facilitating daily patient care and research studies in IBD. This study will focus only on patients with UC enrolled in the UR-CARE platform.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Malignancy excluding non-melanoma skin cancer (NMSC) | from 01 July 2018 through to 31 March 2025
  Malignancy excluding non-melanoma skin cancer (NMSC). As this is a post-authorisation safety study requested by the EMA, the physician is simply asked to report whether such an event has occurred in the patient's life and under what treatment. The study does not aim to measure or clinically qualify this event, which is why nothing more is asked to estimate the incidence rates of the event.
venous thromboembolic events (VTE),(deep venous thrombosis [DVT] and pulmonary embolism [PE]) | from 01 July 2018 through to 31 March 2025
  deep venous thrombosis [DVT] and pulmonary embolism [PE]. As this is a post-authorisation safety study requested by the EMA, the physician is simply asked to report whether such an event has occurred in the patient's life and under what treatment. The study does not aim to measure or clinically qualify this event, which is why nothing more is asked to estimate the incidence rates of the event.

SECONDARY OUTCOMES:
Non melanoma skin cancer (NMSC) | from 01 July 2018 through to 31 March 2025
  Non melanoma skin cancer (NMSC). As this is a post-authorisation safety study requested by the EMA, the physician is simply asked to report whether such an event has occurred in the patient's life and under what treatment. The study does not aim to measure or clinically qualify this event, which is why nothing more is asked to estimate the incidence rates of the event.
Lung cancer | from 01 July 2018 through to 31 March 2025
  Lung cancer. As this is a post-authorisation safety study requested by the EMA, the physician is simply asked to report whether such an event has occurred in the patient's life and under what treatment. The study does not aim to measure or clinically qualify this event, which is why nothing more is asked to estimate the incidence rates of the event.
Lymphoma | from 01 July 2018 through to 31 March 2025
  Lymphoma (including 3 main subtypes Hodgkin's lymphoma, non-Hodgkin's lymphoma, and chronic lymphocytic lymphoma).
  As this is a post-authorisation safety study requested by the EMA, the physician is simply asked to report whether such an event has occurred in the patient's life and under what treatment. The study does not aim to measure or clinically qualify this event, which is why nothing more is asked to estimate the incidence rates of the event.
Serious infections | from 01 July 2018 through to 31 March 2025
  Serious infections. As this is a post-authorisation safety study requested by the EMA, the physician is simply asked to report whether such an event has occurred in the patient's life and under what treatment. The study does not aim to measure or clinically qualify this event, which is why nothing more is asked to estimate the incidence rates of the event.
Opportunistic infections (e.g., tuberculosis) | from 01 July 2018 through to 31 March 2025
  Opportunistic infections (e.g., tuberculosis). As this is a post-authorisation safety study requested by the EMA, the physician is simply asked to report whether such an event has occurred in the patient's life and under what treatment. The study does not aim to measure or clinically qualify this event, which is why nothing more is asked to estimate the incidence rates of the event.
Herpes zoster(HZ) | from 01 July 2018 through to 31 March 2025
  Herpes zoster(HZ). As this is a post-authorisation safety study requested by the EMA, the physician is simply asked to report whether such an event has occurred in the patient's life and under what treatment. The study does not aim to measure or clinically qualify this event, which is why nothing more is asked to estimate the incidence rates of the event.
Major adverse cardiac events (MACE) | from 01 July 2018 through to 31 March 2025
  Major adverse cardiac events (MACE)
Myocardial infarction (MI) | from 01 July 2018 through to 31 March 2025
  Myocardial infarction (MI). As this is a post-authorisation safety study requested by the EMA, the physician is simply asked to report whether such an event has occurred in the patient's life and under what treatment. The study does not aim to measure or clinically qualify this event, which is why nothing more is asked to estimate the incidence rates of the event.
Progressive multifocal leukoencephalopathy (PML) | from 01 July 2018 through to 31 March 2025
  Progressive multifocal leukoencephalopathy (PML). As this is a post-authorisation safety study requested by the EMA, the physician is simply asked to report whether such an event has occurred in the patient's life and under what treatment. The study does not aim to measure or clinically qualify this event, which is why nothing more is asked to estimate the incidence rates of the event.
Gastrointestinal (GI) perforations | from 01 July 2018 through to 31 March 2025
  Gastrointestinal (GI) perforations. As this is a post-authorisation safety study requested by the EMA, the physician is simply asked to report whether such an event has occurred in the patient's life and under what treatment. The study does not aim to measure or clinically qualify this event, which is why nothing more is asked to estimate the incidence rates of the event.
Fractures | from 01 July 2018 through to 31 March 2025
  Fractures. As this is a post-authorisation safety study requested by the EMA, the physician is simply asked to report whether such an event has occurred in the patient's life and under what treatment. The study does not aim to measure or clinically qualify this event, which is why nothing more is asked to estimate the incidence rates of the event.
All-cause mortality | from 01 July 2018 through to 31 March 2025
  All-cause mortality
surgery for Ulcerative colitis (UC) | from 01 July 2018 through to 31 March 2025
  surgery for Ulcerative colitis (UC). As this is a post-authorisation safety study requested by the EMA, the physician is simply asked to report whether such an event has occurred in the patient's life and under what treatment. The study does not aim to measure or clinically qualify this event, which is why nothing more is asked to estimate the incidence rates of the event.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel MD Barreiro, PhD, Principal Investigator — Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa
Locations (5):
- Belgium (2):
  - Imelda General Hospital, Bonheiden
  - AZ Delta vzw, Roeselare
- Acibadem City Clinic Tokuda University Hospital, Sofia, Bulgaria
- General Hospital of Athens "Evangelismos", Ellinikó, Attica, Greece
- Lithuanian University of Life Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burisch J, Pedersen N, Cukovic-Cavka S, Brinar M, Kaimakliotis I, Duricova D, Shonova O, Vind I, Avnstrom S, Thorsgaard N, Andersen V, Krabbe S, Dahlerup JF, Salupere R, Nielsen KR, Olsen J, Manninen P, Collin P, Tsianos EV, Katsanos KH, Ladefoged K, Lakatos L, Bjornsson E, Ragnarsson G, Bailey Y, Odes S, Schwartz D, Martinato M, Lupinacci G, Milla M, De Padova A, D'Inca R, Beltrami M, Kupcinskas L, Kiudelis G, Turcan S, Tighineanu O, Mihu I, Magro F, Barros LF, Goldis A, Lazar D, Belousova E, Nikulina I, Hernandez V, Martinez-Ares D, Almer S, Zhulina Y, Halfvarson J, Arebi N, Sebastian S, Lakatos PL, Langholz E, Munkholm P; EpiCom-group. East-West gradient in the incidence of inflammatory bowel disease in Europe: the ECCO-EpiCom inception cohort. Gut. 2014 Apr;63(4):588-97. doi: 10.1136/gutjnl-2013-304636. Epub 2013 Apr 20. PMID 23604131
- [Background] Sjoberg D, Holmstrom T, Larsson M, Nielsen AL, Holmquist L, Ekbom A, Ronnblom A. Incidence and natural history of ulcerative colitis in the Uppsala Region of Sweden 2005-2009 - results from the IBD cohort of the Uppsala Region (ICURE). J Crohns Colitis. 2013 Oct;7(9):e351-7. doi: 10.1016/j.crohns.2013.02.006. Epub 2013 Mar 9. PMID 23491313
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Busch K, Ludvigsson JF, Ekstrom-Smedby K, Ekbom A, Askling J, Neovius M. Nationwide prevalence of inflammatory bowel disease in Sweden: a population-based register study. Aliment Pharmacol Ther. 2014 Jan;39(1):57-68. doi: 10.1111/apt.12528. Epub 2013 Oct 16. PMID 24127738
- [Background] The Committee for Medicinal Products for Human Use. Guideline on the development of new medicinal products for the treatment of ulcerative colitis. CHMP/EWP/18463/2006 Revision 1. Available at: https://www.ema.europa.eu/en/documents/scientific-guideline/guideline-development-new-medicinal-products-treatment-ulcerative-colitis-revision-1_en.pdf
- [Background] Coward S, Clement F, Benchimol EI, Bernstein CN, Avina-Zubieta JA, Bitton A, Carroll MW, Hazlewood G, Jacobson K, Jelinski S, Deardon R, Jones JL, Kuenzig ME, Leddin D, McBrien KA, Murthy SK, Nguyen GC, Otley AR, Panaccione R, Rezaie A, Rosenfeld G, Pena-Sanchez JN, Singh H, Targownik LE, Kaplan GG. Past and Future Burden of Inflammatory Bowel Diseases Based on Modeling of Population-Based Data. Gastroenterology. 2019 Apr;156(5):1345-1353.e4. doi: 10.1053/j.gastro.2019.01.002. Epub 2019 Jan 10. PMID 30639677
- [Background] Dahlhamer JM, Zammitti EP, Ward BW, Wheaton AG, Croft JB. Prevalence of Inflammatory Bowel Disease Among Adults Aged >/=18 Years - United States, 2015. MMWR Morb Mortal Wkly Rep. 2016 Oct 28;65(42):1166-1169. doi: 10.15585/mmwr.mm6542a3. PMID 27787492
- [Background] Everhov AH, Halfvarson J, Myrelid P, Sachs MC, Nordenvall C, Soderling J, Ekbom A, Neovius M, Ludvigsson JF, Askling J, Olen O. Incidence and Treatment of Patients Diagnosed With Inflammatory Bowel Diseases at 60 Years or Older in Sweden. Gastroenterology. 2018 Feb;154(3):518-528.e15. doi: 10.1053/j.gastro.2017.10.034. Epub 2017 Nov 2. PMID 29102619
- [Background] Khalili, H., Söderling, J., Everhov, Å. H., et al. 15 - Health Care Use, Work Loss, and Total Costs in Incident and Prevelant Ulcerative Colitis: Results from a Nationwide Study in Sweden. Gastroenterology 2018, 154(Supplement 1), S-5-5. http://doi.org/10.1016/S0016-5085(18)30504-3
- [Background] Sandborn WJ, Ghosh S, Panes J, Vranic I, Su C, Rousell S, Niezychowski W; Study A3921063 Investigators. Tofacitinib, an oral Janus kinase inhibitor, in active ulcerative colitis. N Engl J Med. 2012 Aug 16;367(7):616-24. doi: 10.1056/NEJMoa1112168. PMID 22894574
- [Background] Lichtenstein GR, Abreu MT, Cohen R, Tremaine W; American Gastroenterological Association. American Gastroenterological Association Institute technical review on corticosteroids, immunomodulators, and infliximab in inflammatory bowel disease. Gastroenterology. 2006 Mar;130(3):940-87. doi: 10.1053/j.gastro.2006.01.048. No abstract available. PMID 16530532
- [Background] McAuliffe ME, Lanes S, Leach T, Parikh A, Faich G, Porter J, Holick C, Esposito D, Zhao Y, Fox I. Occurrence of adverse events among patients with inflammatory bowel disease in the HealthCore Integrated Research Database. Curr Med Res Opin. 2015;31(9):1655-64. doi: 10.1185/03007995.2015.1065242. Epub 2015 Aug 20. PMID 26135040
- [Background] Ludvigsson JF, Svedberg P, Olen O, Bruze G, Neovius M. The longitudinal integrated database for health insurance and labour market studies (LISA) and its use in medical research. Eur J Epidemiol. 2019 Apr;34(4):423-437. doi: 10.1007/s10654-019-00511-8. Epub 2019 Mar 30. PMID 30929112
- [Background] Biemans VBC, van der Meulen-de Jong AE, van der Woude CJ, Lowenberg M, Dijkstra G, Oldenburg B, de Boer NKH, van der Marel S, Bodelier AGL, Jansen JM, Haans JJL, Theeuwen R, de Jong D, Pierik MJ, Hoentjen F. Ustekinumab for Crohn's Disease: Results of the ICC Registry, a Nationwide Prospective Observational Cohort Study. J Crohns Colitis. 2020 Jan 1;14(1):33-45. doi: 10.1093/ecco-jcc/jjz119. PMID 31219157
- [Background] Zabana Y, Panes J, Nos P, Gomollon F, Esteve M, Garcia-Sanchez V, Gisbert JP, Barreiro-de-Acosta M, Domenech E; en representacion de GETECCU. The ENEIDA registry (Nationwide study on genetic and environmental determinants of inflammatory bowel disease) by GETECCU: Design, monitoring and functions. Gastroenterol Hepatol. 2020 Nov;43(9):551-558. doi: 10.1016/j.gastrohep.2020.05.007. Epub 2020 Jul 14. English, Spanish. PMID 32674882
- [Background] Murthy SK, Robertson McCurdy AB, Carrier M, McCurdy JD. Venous thromboembolic events in inflammatory bowel diseases: A review of current evidence and guidance on risk in the post-hospitalization setting. Thromb Res. 2020 Oct;194:26-32. doi: 10.1016/j.thromres.2020.06.005. Epub 2020 Jun 3. PMID 32563061
- [Background] Curtis JR, Chen SY, Werther W, John A, Johnson DA. Validation of ICD-9-CM codes to identify gastrointestinal perforation events in administrative claims data among hospitalized rheumatoid arthritis patients. Pharmacoepidemiol Drug Saf. 2011 Nov;20(11):1150-8. doi: 10.1002/pds.2215. Epub 2011 Aug 27. PMID 22020901
- [Background] Brooke, H. L., Holzmann, M. J., Olen, O., et al. Enhancing evidence-based medicine: Twelve tips for conducting register-based research. MedEdPublish 2016; 5(2). http://doi.org/10.15694/mep.2016.000071
- [Background] Bernstein CN, Blanchard JF, Kliewer E, Wajda A. Cancer risk in patients with inflammatory bowel disease: a population-based study. Cancer. 2001 Feb 15;91(4):854-62. doi: 10.1002/1097-0142(20010215)91:43.0.co;2-z. PMID 11241255
- [Background] Jess T, Horvath-Puho E, Fallingborg J, Rasmussen HH, Jacobsen BA. Cancer risk in inflammatory bowel disease according to patient phenotype and treatment: a Danish population-based cohort study. Am J Gastroenterol. 2013 Dec;108(12):1869-76. doi: 10.1038/ajg.2013.249. Epub 2013 Aug 27. PMID 23978954
- [Background] van den Heuvel TR, Wintjens DS, Jeuring SF, Wassink MH, Romberg-Camps MJ, Oostenbrug LE, Sanduleanu S, Hameeteman WH, Zeegers MP, Masclee AA, Jonkers DM, Pierik MJ. Inflammatory bowel disease, cancer and medication: Cancer risk in the Dutch population-based IBDSL cohort. Int J Cancer. 2016 Sep 15;139(6):1270-80. doi: 10.1002/ijc.30183. Epub 2016 May 31. PMID 27170593
- [Background] Mercer LK, Lunt M, Low AL, Dixon WG, Watson KD, Symmons DP, Hyrich KL; BSRBR Control Centre Consortium. Risk of solid cancer in patients exposed to anti-tumour necrosis factor therapy: results from the British Society for Rheumatology Biologics Register for Rheumatoid Arthritis. Ann Rheum Dis. 2015 Jun;74(6):1087-93. doi: 10.1136/annrheumdis-2013-204851. Epub 2014 Mar 31. PMID 24685910
- [Background] Mercer LK, Galloway JB, Lunt M, Davies R, Low AL, Dixon WG, Watson KD; BSRBR Control Centre Consortium; Symmons DP, Hyrich KL. Risk of lymphoma in patients exposed to antitumour necrosis factor therapy: results from the British Society for Rheumatology Biologics Register for Rheumatoid Arthritis. Ann Rheum Dis. 2017 Mar;76(3):497-503. doi: 10.1136/annrheumdis-2016-209389. Epub 2016 Aug 8. PMID 27502891
- [Background] Strangfeld A, Hierse F, Rau R, Burmester GR, Krummel-Lorenz B, Demary W, Listing J, Zink A. Risk of incident or recurrent malignancies among patients with rheumatoid arthritis exposed to biologic therapy in the German biologics register RABBIT. Arthritis Res Ther. 2010;12(1):R5. doi: 10.1186/ar2904. Epub 2010 Jan 8. PMID 20064207
- [Background] Wadstrom H, Frisell T, Askling J; Anti-Rheumatic Therapy in Sweden (ARTIS) Study Group. Malignant Neoplasms in Patients With Rheumatoid Arthritis Treated With Tumor Necrosis Factor Inhibitors, Tocilizumab, Abatacept, or Rituximab in Clinical Practice: A Nationwide Cohort Study From Sweden. JAMA Intern Med. 2017 Nov 1;177(11):1605-1612. doi: 10.1001/jamainternmed.2017.4332. PMID 28975211
- [Background] Ludvigsson JF, Andersson M, Bengtsson J, Eberhardson M, Fagerberg UL, Grip O, Halfvarson J, Hjortswang H, Jaghult S, Karling P, Nordenvall C, Olen O, Olsson M, Rejler M, Strid H, Myrelid P. Swedish Inflammatory Bowel Disease Register (SWIBREG) - a nationwide quality register. Scand J Gastroenterol. 2019 Sep;54(9):1089-1101. doi: 10.1080/00365521.2019.1660799. Epub 2019 Sep 9. PMID 31498717
- [Background] Abdul Sultan A, West J, Stephansson O, Grainge MJ, Tata LJ, Fleming KM, Humes D, Ludvigsson JF. Defining venous thromboembolism and measuring its incidence using Swedish health registries: a nationwide pregnancy cohort study. BMJ Open. 2015 Nov 11;5(11):e008864. doi: 10.1136/bmjopen-2015-008864. PMID 26560059
- [Background] Degli Esposti L, Favalli EG, Sangiorgi D, Di Turi R, Farina G, Gambera M, Ravasio R. Persistence, switch rates, drug consumption and costs of biological treatment of rheumatoid arthritis: an observational study in Italy. Clinicoecon Outcomes Res. 2016 Dec 21;9:9-17. doi: 10.2147/CEOR.S108730. eCollection 2017. PMID 28053549
- [Background] Chaparro M, Ramas M, Benitez JM, Lopez-Garcia A, Juan A, Guardiola J, Minguez M, Calvet X, Marquez L, Fernandez Salazar LI, Bujanda L, Garcia C, Zabana Y, Lorente R, Barrio J, Hinojosa E, Iborra M, Cajal MD, Van Domselaar M, Garcia-Sepulcre MF, Gomollon F, Piqueras M, Alcain G, Garcia-Sanchez V, Panes J, Domenech E, Garcia-Esquinas E, Rodriguez-Artalejo F, Gisbert JP. Extracolonic Cancer in Inflammatory Bowel Disease: Data from the GETECCU Eneida Registry. Am J Gastroenterol. 2017 Jul;112(7):1135-1143. doi: 10.1038/ajg.2017.96. Epub 2017 May 23. PMID 28534520
- [Background] Scharl S, Barthel C, Rossel JB, Biedermann L, Misselwitz B, Schoepfer AM, Straumann A, Vavricka SR, Rogler G, Scharl M, Greuter T. Malignancies in Inflammatory Bowel Disease: Frequency, Incidence and Risk Factors-Results from the Swiss IBD Cohort Study. Am J Gastroenterol. 2019 Jan;114(1):116-126. doi: 10.1038/s41395-018-0360-9. PMID 30333538
- [Background] Papa A, Gerardi V, Marzo M, Felice C, Rapaccini GL, Gasbarrini A. Venous thromboembolism in patients with inflammatory bowel disease: focus on prevention and treatment. World J Gastroenterol. 2014 Mar 28;20(12):3173-9. doi: 10.3748/wjg.v20.i12.3173. PMID 24695669